CLINICAL TRIAL: NCT02061683
Title: A Study of Bimatoprost in the Treatment of Primary Open Angle Glaucoma and Ocular Hypertension
Acronym: LOTUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN-BIM-0901
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bimatoprost 0.03% (Experimental): Bimatoprost 0.03% (LUMIGAN®) 1 drop in the affected eye(s) once daily as monotherapy or adjunctive therapy for 3 months.
  Interventions: Drug: Bimatoprost 0.03%

INTERVENTIONS:
Drug: Bimatoprost 0.03% — Bimatoprost 0.03% (LUMIGAN®) 1 drop in the affected eye(s) once daily as monotherapy or adjunctive therapy for 3 months.
  Other Names: LUMIGAN®

SUMMARY:
This is a study of bimatoprost as initial, replacement, or adjunctive intraocular pressure (IOP)-lowering therapy in patients with primary open angle glaucoma and ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension
* No use of Lumigan® in the past 3 months

Exclusion Criteria:

* Received laser therapy, glaucoma surgery, cataract surgery, or other ocular surgery within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2010-04-19 (Actual); Primary Completion 2011-06-24 (Actual); Study Completion 2011-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Shanghai, China

REFERENCES:
- [Background] Wang K, Xu L, Yuan Z, Yao K, Zhao J, Xu L, Fang A, Zhang M, Wu L, Ji J, Hou J, Liu Q, Sun X. Intraocular pressure-lowering efficacy and safety of bimatoprost 0.03% therapy for primary open-angle glaucoma and ocular hypertension patients in China. BMC Ophthalmol. 2014 Feb 25;14:21. doi: 10.1186/1471-2415-14-21. PMID 24568617

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost 0.03%
Started | 263
Completed | 203
Not Completed | 60

BASELINE CHARACTERISTICS:
Arm/Group | Bimatoprost 0.03%
Number analyzed (Participants) | 263
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.7 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 155

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) in the Study Eye
Description: IOP is a measure of the fluid pressure inside the study eye. Patients were categorized by pre-study therapies and the bimatoprost-containing study therapy into the following 5 groups: Group A (pre-study: treatment naïve; during study: bimatoprost monotherapy); Group B (pre-study: prostaglandin analog [PGA] monotherapy, excluding bimatoprost; during study: bimatoprost monotherapy); Group C (pre-study: non-PGA monotherapy or combination therapy; during study: bimatoprost monotherapy); Group D (pre-study: combination therapy including PGA, without bimatoprost; during study: pre-study combination therapy with PGA switched to bimatoprost); and Group E (pre-study: non-PGA monotherapy or combination therapy; during study: bimatoprost adjunctive to pre-study therapy).
Time Frame: Month 3
Population: All enrolled patients with data available for analysis
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.03%
Number analyzed (Participants) | 240
Millimeters of Mercury (mmHg)
  Group A (N=89) | 16.5 (3.4)
  Group B (N=33) | 16.7 (3.3)
  Group C (N=67) | 15.7 (2.6)
  Group D (N=18) | 16.1 (3.5)
  Group E (N=33) | 17.2 (4.4)

2. Secondary Outcome: Percentage of Patients With an Adverse Event of Conjunctival Hyperemia
Description: Conjunctival hyperemia is engorgement of the blood vessels (redness) of the bulbar conjunctiva of the eye (the clear membrane covering the white surface of the eye). An adverse event is any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug.
Time Frame: 3 Months
Population: Safety population defined as all enrolled patients who completed at least 1 follow-up visit
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost 0.03%
Number analyzed (Participants) | 250
Percentage of Patients | 76.0

ADVERSE EVENTS:
Description: The safety population was used to assess adverse events (AEs) and serious adverse events (SAEs), and was defined as all enrolled patients who completed at least 1 follow-up visit.
Arm/Group | Bimatoprost 0.03%
Serious Adverse Events (participants affected / at risk) | 0/250
Other Adverse Events (participants affected / at risk) | 229/250
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.03% (N=250)
Eyelash growth (Eye disorders) | 23
Skin pigmentation (Skin and subcutaneous tissue disorders) | 16
Conjunctival Hyperemia (Eye disorders) | 190

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of at least 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.